CLINICAL TRIAL: NCT05827068
Title: A Phase 1/2, Randomized, Open-Label Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of mRNA-1011.1, mRNA-1011.2, and mRNA-1012.1 Candidate Seasonal Influenza Vaccines in Healthy Adults 50 to 75 Years of Age
Brief Title: A Study of mRNA-1011.1, mRNA-1011.2, and mRNA-1012.1 Candidate Seasonal Influenza Vaccines in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: mRNA-1011-P101
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Seasonal Influenza
Keywords: Influenza vaccine; mRNA-1010; mRNA-1011.1; mRNA-1011.2; mRNA-1012.1; Moderna
MeSH Terms: conditions — Influenza, Human | interventions — mRNA-1010 influenza vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- mRNA-1011.1 (Experimental): Participants will receive mRNA-1011.1 by intramuscular (IM) injection on Day 1.
  Interventions: Biological: mRNA-1011.1
- mRNA-1011.2 (Experimental): Participants will receive mRNA-1011.2 by IM injection on Day 1.
  Interventions: Biological: mRNA-1011.2
- mRNA-1012.1 Dose Level A (Experimental): Participants will receive mRNA-1012.1 at dose level A by IM injection on Day 1.
  Interventions: Biological: mRNA-1012.1
- mRNA-1012.1 Dose Level B (Experimental): Participants will receive mRNA-1012.1 at dose level B by IM injection on Day 1.
  Interventions: Biological: mRNA-1012.1
- mRNA-1010 (Active Comparator): Participants will receive mRNA-1010 by IM injection on Day 1.
  Interventions: Biological: mRNA-1010
- mRNA-1010.2 (Active Comparator): Participants will receive mRNA-1010.2 by IM injection on Day 1.
  Interventions: Biological: mRNA-1010.2
- mRNA-1010.3 (Active Comparator): Participants will receive mRNA-1010.3 by IM injection on Day 1.
  Interventions: Biological: mRNA-1010.3

INTERVENTIONS:
Biological: mRNA-1011.1 — Sterile liquid for injection
  Other Names: Seasonal influenza vaccine
  Arms: mRNA-1011.1
Biological: mRNA-1011.2 — Sterile liquid for injection
  Other Names: Seasonal influenza vaccine
  Arms: mRNA-1011.2
Biological: mRNA-1012.1 — Sterile liquid for injection
  Other Names: Seasonal influenza vaccine
  Arms: mRNA-1012.1 Dose Level A; mRNA-1012.1 Dose Level B
Biological: mRNA-1010 — Sterile liquid for injection
  Other Names: Seasonal influenza vaccine
  Arms: mRNA-1010
Biological: mRNA-1010.2 — Sterile liquid for injection
  Other Names: Seasonal influenza vaccine
  Arms: mRNA-1010.2
Biological: mRNA-1010.3 — Sterile liquid for injection
  Other Names: Seasonal influenza vaccine
  Arms: mRNA-1010.3

SUMMARY:
The purpose of this study is to measure the safety and the immune response to 3 next-generation influenza vaccine candidates (mRNA-1011.1, mRNA-1011.2, and mRNA-1012.1) compared with influenza vaccine candidate mRNA-1010 controls in healthy adult participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index of 18 kilograms (kg)/square meter (m^2) to 35 kg/m^2 (inclusive) at the Screening Visit.
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1, agreement to continue adequate contraception through 3 months following vaccine administration, and not currently breastfeeding.

Key Exclusion Criteria:

* Participant is acutely ill or febrile (temperature ≥38.0 degrees Celsius [°C]/100.4 degrees Fahrenheit [°F]) 72 hours prior to or at the Screening Visit or Day 1.
* Any medical, psychiatric, or occupational condition, including reported history of substance abuse, that, in the opinion of the Investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.
* Participant has received systemic immunosuppressants for >14 days in total within 180 days prior to the Randomization Visit (for glucocorticosteroids ≥10 milligrams [mg]/day of prednisone equivalent) or is anticipating the need for systemic immunosuppressive treatment at any time during participation in the study (including intra-articular steroid injections). Inhaled, nasal, and topical steroids are allowed.
* Participant has received or plans to receive any licensed or authorized vaccine, including COVID-19 vaccines, ≤28 days prior to the study injection (Day 1) or plans to receive a licensed or authorized vaccine within 28 days after the study injection.
* Participant has received a seasonal influenza vaccine or any other influenza vaccine within 180 days prior to the Randomization Visit.
* Participant tested positive for influenza by local health authority-approved testing methods within 180 days prior to the Randomization Visit.
* Participant has had close contact to someone with or been diagnosed themselves with respiratory syncytial virus or SARS-CoV-2 infection as defined by the Centers for Disease Control and Prevention (CDC) in the past 10 days prior to the Randomization Visit.
* Participant has donated ≥450 milliliters (mL) of blood products within 28 days prior to the Randomization Visit or plans to donate blood products during the study.

Note: Other inclusion/exclusion criteria may apply.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Long Beach Research Institute, Lakewood, California
  - Long Beach Clinical Trials, Long Beach, California
  - Tekton Research, Fort Collins, Colorado
  - Critical Care, Pulmonary and Sleep Associates / CCT Research, Lakewood, Colorado
  - CenExel RCA, Hollywood, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - CenExel FCR, Tampa, Florida
  - Georgia Clinic / CCT Research, Norcross, Georgia
  - CenExel CBH, Gaithersburg, Maryland
  - DelRicht Research, Rockville, Maryland
  - DelRicht Research, Springfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - DelRicht Research, Town and Country, Missouri
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Healor Primary Care, Las Vegas, Nevada
  - Meridian Clinical Research, LLC, Vestal, New York
  - Tekton Research, Edmond, Oklahoma
  - Tekton Research, Moore, Oklahoma
  - The Corvallis Clinic, PC, Corvallis, Oregon
  - Hatboro Medical Associates / CCT Research, Hatboro, Pennsylvania
  - Trial Management Associates, LLC, Myrtle Beach, South Carolina
  - Springville Dermatology / CCT Research, Springville, Utah

REFERENCES:
- [Derived] Hsu D, Jayaraman A, Pucci A, Joshi R, Mancini K, Chen HL, Koslovsky K, Mao X, Choi A, Henry C, Vakil J, Stadlbauer D, Jorquera P, Arunkumar GA, Sanchez-Crespo NE, Wadsworth LT, Bhupathy V, Du E, Avanesov A, Ananworanich J, Nachbagauer R. Safety and immunogenicity of mRNA-based seasonal influenza vaccines formulated to include multiple A/H3N2 strains with or without the B/Yamagata strain in US adults aged 50-75 years: a phase 1/2, open-label, randomised trial. Lancet Infect Dis. 2025 Jan;25(1):25-35. doi: 10.1016/S1473-3099(24)00493-6. Epub 2024 Sep 5. PMID 39245055

RESULTS

PARTICIPANT FLOW:
Groups:
- mRNA-1010 50 μg: Participants received a single intramuscular (IM) injection of mRNA-1010 50 micrograms (μg) on Day 1.
- mRNA-1010.2 50 μg: Participants received a single IM injection of mRNA-1010.2 50 μg on Day 1.
- mRNA-1010.3 50 μg: Participants received a single IM injection of mRNA-1010.3 50 μg on Day 1.
- mRNA-1011.1 50 μg: Participants received a single IM injection of mRNA-1011.1 50 μg on Day 1.
- mRNA-1011.2 40 μg: Participants received a single IM injection of mRNA-1011.2 40 μg on Day 1.
- mRNA-1012.1 50 μg: Participants received a single IM injection of mRNA-1012.1 50 μg on Day 1.
- mRNA-1012.1 62.5 μg: Participants received a single IM injection of mRNA-1012.1 62.5 μg on Day 1.
Period: Overall Study
Arm/Group | mRNA-1010 50 μg | mRNA-1010.2 50 μg | mRNA-1010.3 50 μg | mRNA-1011.1 50 μg | mRNA-1011.2 40 μg | mRNA-1012.1 50 μg | mRNA-1012.1 62.5 μg
Started (Randomized Participants) | 99 | 101 | 98 | 99 | 100 | 100 | 101
Received Injection | 99 | 100 | 97 | 99 | 100 | 100 | 100
Safety Set (All randomly assigned participants who received the study vaccination.) | 99 | 100 | 97 | 99 | 100 | 100 | 98
Solicited Safety Set (All randomly assigned participants who received the study vaccination and contributed any solicited AR data.) | 99 | 100 | 97 | 98 | 100 | 100 | 97
Participants Were Randomized to mRNA-1012.1 62.5 μg But Received mRNA-1012.1 50 μg Instead (These 2 participants were included in mRNA-1012.1 50 μg group for Safety Set and Solicited Safety Set.) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2 Participants randomized to receive mRNA-1012.1 62.5 μg but actually received mRNA-1012.1 50 μg.)
Completed | 94 | 96 | 96 | 96 | 94 | 96 | 98
Not Completed | 5 | 5 | 2 | 3 | 6 | 4 | 3
Not completed — Lost to Follow-up | 1 | 4 | 1 | 1 | 2 | 4 | 1
Not completed — Withdrawal by Subject | 4 | 0 | 1 | 2 | 3 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Other Than Specified | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all randomly assigned participants who received the study vaccination.
Groups:
- mRNA-1010 50 μg: Participants received a single IM injection of mRNA-1010 50 μg on Day 1.
- Total: Total of all reporting groups
Arm/Group | mRNA-1010 50 μg | mRNA-1010.2 50 μg | mRNA-1010.3 50 μg | mRNA-1011.1 50 μg | mRNA-1011.2 40 μg | mRNA-1012.1 50 μg | mRNA-1012.1 62.5 μg | Total
Number analyzed (Participants) | 99 | 100 | 97 | 99 | 100 | 100 | 100 | 695
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (7.17) | 62.2 (6.95) | 60.8 (7.47) | 61.4 (6.17) | 61.6 (7.18) | 60.7 (7.79) | 61.1 (6.70) | 61.2 (7.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 62 | 53 | 52 | 61 | 48 | 53 | 381
  Male | 47 | 38 | 44 | 47 | 39 | 52 | 47 | 314
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 20 | 12 | 21 | 25 | 20 | 19 | 138
  Not Hispanic or Latino | 77 | 75 | 84 | 76 | 72 | 77 | 81 | 542
  Unknown or Not Reported | 1 | 5 | 1 | 2 | 3 | 3 | 0 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 1 | 2 | 1 | 1 | 0 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Black or African American | 10 | 22 | 20 | 23 | 13 | 13 | 21 | 122
  White | 86 | 75 | 74 | 72 | 84 | 86 | 75 | 552
  More than one race | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 2 | 1 | 0 | 2 | 0 | 1 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs)
Description: Solicited ARs (local and systemic) were collected in an electronic diary (eDiary). Local ARs included: injection site pain, injection site erythema (redness), injection site swelling/induration (hardness), and axillary (underarm) swelling or tenderness ipsilateral to the side of injection. Systemic ARs included: fever, headache, fatigue, myalgia, arthralgia, nausea/vomiting, and chills. All solicited ARs considered causally related to injection were graded 0-4 (per Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials); lower score indicates lower severity, and a higher score indicates greater severity.
Time Frame: 7 days post-vaccination
Population: The Solicited Safety Set included all randomly assigned participants who received the study vaccination and contributed any solicited AR data. Participants were included in the vaccination group corresponding to what they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1010 50 μg | mRNA-1010.2 50 μg | mRNA-1010.3 50 μg | mRNA-1011.1 50 μg | mRNA-1011.2 40 μg | mRNA-1012.1 50 μg | mRNA-1012.1 62.5 μg
Number analyzed (Participants) | 99 | 100 | 97 | 98 | 100 | 102 | 97
Participants
  Any | 77 | 86 | 81 | 72 | 75 | 85 | 74
  Grade 1 | 42 | 45 | 31 | 29 | 41 | 40 | 33
  Grade 2 | 30 | 38 | 43 | 37 | 30 | 37 | 38
  Grade 3 | 5 | 3 | 7 | 6 | 4 | 8 | 3
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Unsolicited AEs
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Any abnormal laboratory test result (hematology, clinical chemistry, or prothrombin time [PT]/partial thromboplastin time [PTT]) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsened from baseline and was considered clinically significant in the medical and scientific judgment of the Investigator was recorded as an AE. Number of participants with unsolicited AEs (SAEs and non-serious AEs) up to 28 days post-vaccination are reported in this outcome measure.
Time Frame: Up to 28 days post-vaccination
Population: The Safety Set included all randomly assigned participants who received the study vaccination. Participants were included in the vaccination group corresponding to what they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1010 50 μg | mRNA-1010.2 50 μg | mRNA-1010.3 50 μg | mRNA-1011.1 50 μg | mRNA-1011.2 40 μg | mRNA-1012.1 50 μg | mRNA-1012.1 62.5 μg
Number analyzed (Participants) | 99 | 100 | 97 | 99 | 100 | 102 | 98
Participants | 11 | 17 | 15 | 6 | 7 | 10 | 16

3. Primary Outcome: Number of Participants With SAEs, AEs of Special Interest (AESIs), Medically Attended AEs (MAAEs), and AEs Leading to Discontinuation
Description: An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. AESIs included thrombocytopenia, new onset of or worsening of the protocol specified neurologic diseases, anaphylaxis, and myocarditis/pericarditis. An MAAE is an AE that lead to an unscheduled visit to an healthcare practitioner. This included visits to a study site for unscheduled assessments (for example, abnormal laboratory follow-up) and visits to healthcare practitioners external to the study site (for example, urgent care, primary care physician). Number of participants with SAEs, AESIs, MAAEs, and AEs leading to discontinuation up to the end of study (Day 181) are reported in this outcome measure.
Time Frame: Day 1 to Day 181 (end of study [EOS])
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | mRNA-1010 50 μg | mRNA-1010.2 50 μg | mRNA-1010.3 50 μg | mRNA-1011.1 50 μg | mRNA-1011.2 40 μg | mRNA-1012.1 50 μg | mRNA-1012.1 62.5 μg
Number analyzed (Participants) | 99 | 100 | 97 | 99 | 100 | 102 | 98
Participants
  SAEs | 2 | 3 | 1 | 0 | 2 | 2 | 3
  AESIs | 0 | 0 | 0 | 0 | 0 | 1 | 1
  MAAEs | 10 | 21 | 18 | 12 | 24 | 23 | 16
  AEs Leading to Discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Geometric Mean Titer (GMT) of Anti-Hemagglutinin (HA) Antibodies at Day 29, as Measured by Hemagglutination Inhibition (HAI) Assay for Vaccine-matched Influenza A and B Strains
Description: Seasonal influenza A strains included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage.
Time Frame: Day 29
Population: Per-Protocol (PP) Set included all randomly assigned participants who received study vaccination, complied with the injection schedule, complied with the timings of immunogenicity blood sampling to have a baseline and at least the Day 29 post-injection assessment, had no RT-PCR-confirmed influenza infection prior to Day 29 visit and had no major protocol deviations that impacted the immune response. Participants were analyzed according to the group to which they were randomized.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | mRNA-1010 50 μg | mRNA-1010.2 50 μg | mRNA-1010.3 50 μg | mRNA-1011.1 50 μg | mRNA-1011.2 40 μg | mRNA-1012.1 50 μg | mRNA-1012.1 62.5 μg
Number analyzed (Participants) | 93 | 89 | 95 | 87 | 90 | 92 | 88
titer
  Influenza A H1N1 Antibody | 197.9 [156.37 to 250.35] | 214.3 [174.66 to 262.85] | 204.3 [163.67 to 255.05] | 189.1 [149.05 to 239.98] | 207.2 [165.10 to 259.97] | 188.9 [154.11 to 231.47] | 216.7 [174.91 to 268.52]
  Influenza A H3N2 (Darwin) Antibody | 122.3 [99.84 to 149.93] | 79.4 [63.87 to 98.62] | 83.3 [69.50 to 99.76] | 117.8 [95.33 to 145.44] | 138.2 [108.34 to 176.27] | 115.7 [94.61 to 141.59] | 122.0 [98.63 to 150.86]
  Influenza A H3N2 (Newcastle) Antibody | 130.8 [104.44 to 163.90] | 205.3 [168.20 to 250.58] | 127.2 [106.29 to 152.10] | 178.2 [142.20 to 223.29] | 232.2 [188.10 to 286.53] | 187.4 [151.33 to 232.06] | 224.5 [179.54 to 280.60]
  Influenza A H3N2 (Hong Kong) Antibody | 73.4 [59.36 to 90.80] | 82.2 [67.36 to 100.33] | 97.1 [82.28 to 114.53] | 86.9 [68.07 to 111.03] | 111.8 [90.22 to 138.50] | 105.0 [85.77 to 128.43] | 122.9 [99.89 to 151.25]
  Influenza B/ Yamagata Lineage | 111.1 [98.52 to 125.25] | 125.2 [106.42 to 147.30] | 118.7 [103.20 to 136.49] | 113.2 [97.59 to 131.32] | 81.6 [71.33 to 93.38] | 77.1 [67.58 to 87.88] | 71.7 [64.20 to 80.00]
  Influenza B/ Victoria Lineage | 207.7 [179.36 to 240.54] | 234.4 [198.48 to 276.72] | 192.0 [162.22 to 227.25] | 197.7 [167.69 to 232.97] | 209.5 [174.89 to 250.88] | 204.4 [172.26 to 242.52] | 211.6 [182.90 to 244.86]

5. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Anti-HA Antibodies at Day 29, as Measured by HAI Assay for Vaccine-matched Influenza A and B Strains
Description: The GMFR measures the changes in immunogenicity titers or levels from Baseline within participants. Seasonal influenza A included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage. Fold-rise was calculated by dividing post-vaccination results by the baseline value. 95% confidence interval (CI) for GMFR was calculated based on the t distribution of the differences in the log-transformed values between analysis timepoint and baseline, then back transformed to the original scale for presentation.
Time Frame: Baseline, Day 29
Population: The PP Set included all randomly assigned participants who received study vaccination, complied with the injection schedule, complied with the timings of immunogenicity blood sampling to have a baseline and at least the Day 29 post-injection assessment, had no RT-PCR-confirmed influenza infection prior to Day 29 visit and had no major protocol deviations that impacted the immune response. Participants were analyzed according to the group to which they were randomized.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | mRNA-1010 50 μg | mRNA-1010.2 50 μg | mRNA-1010.3 50 μg | mRNA-1011.1 50 μg | mRNA-1011.2 40 μg | mRNA-1012.1 50 μg | mRNA-1012.1 62.5 μg
Number analyzed (Participants) | 93 | 89 | 95 | 87 | 90 | 92 | 88
ratio
  Influenza A H1N1 Antibody | 3.0 [2.44 to 3.67] | 3.7 [2.93 to 4.68] | 3.4 [2.86 to 4.16] | 2.7 [2.26 to 3.19] | 3.2 [2.55 to 3.96] | 3.1 [2.59 to 3.82] | 2.9 [2.37 to 3.44]
  Influenza A H3N2 (Darwin) Antibody | 2.8 [2.32 to 3.46] | 2.0 [1.76 to 2.35] | 2.0 [1.77 to 2.31] | 3.1 [2.64 to 3.71] | 3.4 [2.74 to 4.13] | 3.4 [2.88 to 4.08] | 2.6 [2.23 to 3.14]
  Influenza A H3N2 (Newcastle) Antibody | 2.2 [1.79 to 2.78] | 4.0 [3.24 to 4.87] | 2.4 [2.05 to 2.92] | 3.2 [2.66 to 3.86] | 4.2 [3.35 to 5.24] | 4.4 [3.58 to 5.53] | 3.7 [3.00 to 4.59]
  Influenza A H3N2 (Hong Kong) Antibody | 2.7 [2.13 to 3.31] | 3.0 [2.50 to 3.54] | 3.4 [2.87 to 4.08] | 3.1 [2.56 to 3.72] | 4.0 [3.23 to 4.84] | 5.0 [4.10 to 6.14] | 4.1 [3.26 to 5.07]
  Influenza B/Yamagata Lineage | 1.6 [1.41 to 1.80] | 1.9 [1.62 to 2.15] | 1.7 [1.52 to 1.81] | 1.7 [1.50 to 1.86] | 1.2 [1.07 to 1.28] | 1.1 [1.04 to 1.21] | 1.1 [0.99 to 1.13]
  Influenza B/Victoria Lineage | 1.6 [1.36 to 1.81] | 1.8 [1.55 to 2.06] | 1.4 [1.30 to 1.59] | 1.6 [1.44 to 1.78] | 1.8 [1.56 to 2.13] | 1.7 [1.45 to 1.88] | 1.5 [1.34 to 1.72]

6. Secondary Outcome: Percentage of Participants Reaching Seroconversion at Day 29, as Measured by HAI Assay for Vaccine-matched Influenza A and B Strains
Description: Seasonal influenza A strains included H1N1 and H3N2 and seasonal influenza B strains included Victoria-lineage and Yamagata-lineage.
  Seroconversion was defined as a postbaseline titer ≥1:40 if baseline is <1:10 or a 4-fold or greater rise if baseline is ≥1:10 in anti-HA antibodies measured by HAI assay.
Time Frame: Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | mRNA-1010 50 μg | mRNA-1010.2 50 μg | mRNA-1010.3 50 μg | mRNA-1011.1 50 μg | mRNA-1011.2 40 μg | mRNA-1012.1 50 μg | mRNA-1012.1 62.5 μg
Number analyzed (Participants) | 93 | 89 | 95 | 87 | 90 | 92 | 88
percentage of participants
  Influenza A H1N1 Antibody | 36.6 [26.81 to 47.19] | 49.4 [38.67 to 60.25] | 44.2 [34.02 to 54.77] | 40.2 [29.85 to 51.29] | 40.0 [29.81 to 50.87] | 35.9 [26.13 to 46.54] | 35.2 [25.34 to 46.14]
  Influenza A H3N2 (Darwin) Antibody | 40.9 [30.77 to 51.54] | 21.3 [13.37 to 31.31] | 21.1 [13.36 to 30.62] | 40.2 [29.85 to 51.29] | 37.8 [27.77 to 48.62] | 45.7 [35.22 to 56.37] | 33.0 [23.30 to 43.79]
  Influenza A H3N2 (Newcastle) Antibody | 24.7 [16.37 to 34.76] | 53.9 [43.04 to 64.56] | 32.6 [23.36 to 43.02] | 47.1 [36.33 to 58.13] | 52.2 [41.43 to 62.87] | 55.4 [44.70 to 65.81] | 48.9 [38.05 to 59.75]
  Influenza A H3N2 (Hong Kong) Antibody | 34.4 [24.86 to 44.98] | 39.3 [29.13 to 50.25] | 47.4 [37.03 to 57.88] | 44.8 [34.15 to 55.87] | 53.3 [42.51 to 63.93] | 57.6 [46.86 to 67.85] | 52.3 [41.35 to 63.04]
  Influenza B/Yamagata Lineage | 12.9 [6.85 to 21.45] | 16.9 [9.75 to 26.27] | 8.4 [3.71 to 15.92] | 10.3 [4.84 to 18.73] | 1.1 [0.03 to 6.04] | 1.1 [0.03 to 5.91] | 0 [0.00 to 4.11]
  Influenza B/ Victoria Lineage | 10.8 [5.28 to 18.89] | 22.5 [14.30 to 32.55] | 6.3 [2.35 to 13.24] | 9.2 [4.05 to 17.32] | 14.4 [7.92 to 23.43] | 14.1 [7.74 to 22.95] | 11.4 [5.59 to 19.91]

ADVERSE EVENTS:
Time Frame: Day 1 up to the end of study (Day 181)
Description: The all-cause mortality was based on the randomization set. The serious and other (not including serious) adverse events were based on the safety set which consisted of all participants who received one dose of study vaccination. Participants were included in the vaccination group corresponding to what they actually received.
Groups:
- mRNA-1010 50 ug: Participants received a single IM injection of mRNA-1010 50 μg on Day 1.
- mRNA-1010.2 50 ug: Participants received a single IM injection of mRNA-1010.2 50 μg on Day 1.
- mRNA-1010.3 50 ug: Participants received a single IM injection of mRNA-1010.3 50 μg on Day 1.
- mRNA-1011.1 50 ug: Participants received a single IM injection of mRNA-1011.1 50 μg on Day 1.
- mRNA-1011.2 40 ug: Participants received a single IM injection of mRNA-1011.2 40 μg on Day 1.
- mRNA-1012.1 50 ug: Participants received a single IM injection of mRNA-1012.1 50 μg on Day 1.
- mRNA-1012.1 62.5 ug: Participants received a single IM injection of mRNA-1012.1 62.5 μg on Day 1.
Arm/Group | mRNA-1010 50 ug | mRNA-1010.2 50 ug | mRNA-1010.3 50 ug | mRNA-1011.1 50 ug | mRNA-1011.2 40 ug | mRNA-1012.1 50 ug | mRNA-1012.1 62.5 ug
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/101 | 0/98 | 0/99 | 0/100 | 0/100 | 0/101
Serious Adverse Events (participants affected / at risk) | 2/99 | 3/100 | 1/97 | 0/99 | 2/100 | 2/102 | 3/98
Other Adverse Events (participants affected / at risk) | 2/99 | 6/100 | 1/97 | 0/99 | 6/100 | 1/102 | 1/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mRNA-1010 50 ug (N=99) | mRNA-1010.2 50 ug (N=100) | mRNA-1010.3 50 ug (N=97) | mRNA-1011.1 50 ug (N=99) | mRNA-1011.2 40 ug (N=100) | mRNA-1012.1 50 ug (N=102) | mRNA-1012.1 62.5 ug (N=98)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve prolapse (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mRNA-1010 50 ug (N=99) | mRNA-1010.2 50 ug (N=100) | mRNA-1010.3 50 ug (N=97) | mRNA-1011.1 50 ug (N=99) | mRNA-1011.2 40 ug (N=100) | mRNA-1012.1 50 ug (N=102) | mRNA-1012.1 62.5 ug (N=98)
COVID-19 (Infections and infestations) | 2 (2) | 6 (6) | 1 (1) | 0 (0) | 6 (6) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT05827068/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT05827068/SAP_001.pdf